CLINICAL TRIAL: NCT00728949
Title: Phase 2 Randomized, Multicenter Study of IMC-A12 as a Single Agent or in Combination With Antiestrogens in Postmenopausal Women With Hormone Receptor-Positive Advanced or Metastatic Breast Cancer After Progression on Antiestrogen Therapy
Brief Title: A Study for Safety and Effectiveness of IMC-A12 by Itself or Combined With Antiestrogens to Treat Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13935; CP13-0604 (Other: ImClone, LLC); I5A-IE-JAEK (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-07-31; First posted 2008-08-06 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; Postmenopausal; Hormones; Antiestrogen
MeSH Terms: conditions — Breast Neoplasms | interventions — cixutumumab; Tamoxifen; Anastrozole; Letrozole; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMC-A12 (cixutumumab) + antiestrogen therapy (Active Comparator): Participants will receive intravenous IMC-A12 10 mg/kg over 1 hour every 2 weeks, as well as the same dose and schedule of the last antiestrogen therapy to which their disease became refractory.
  Interventions: Biological: IMC-A12 (cixutumumab); Drug: tamoxifen; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant
- IMC-A12 (cixutumumab) (Experimental): Participants will receive only IMC-A12 (10 mg/kg over 1 hour every 2 weeks).
  Interventions: Biological: IMC-A12 (cixutumumab)

INTERVENTIONS:
Biological: IMC-A12 (cixutumumab) — 10 mg/kg I.V.
  Other Names: Cixutumumab; LY3012217
Drug: tamoxifen — Daily 20 mg, oral
  Arms: IMC-A12 (cixutumumab) + antiestrogen therapy
Drug: Anastrozole — Daily 1 mg, oral
  Arms: IMC-A12 (cixutumumab) + antiestrogen therapy
Drug: Letrozole — Daily 2.5 mg, oral
  Arms: IMC-A12 (cixutumumab) + antiestrogen therapy
Drug: Exemestane — Daily 25 mg, oral
  Arms: IMC-A12 (cixutumumab) + antiestrogen therapy
Drug: Fulvestrant — Monthly 250 mg, intramuscularly
  Arms: IMC-A12 (cixutumumab) + antiestrogen therapy

SUMMARY:
The purpose of this study is to determine whether IMC-A12 offers increased progression-free survival (PFS) associated with IMC-A12 monotherapy and IMC-A12 in combination with an antiestrogen therapy in patients with hormone receptor positive advanced or metastatic breast cancer that have experienced disease progression on antiestrogen therapy.

DETAILED DESCRIPTION:
Breast cancer is the most common form of malignancy affecting women worldwide, with approximately 178,480 new cases of invasive breast cancer and 62,030 new cases of in situ breast cancer expected in the United States (US) in 2007. Approximately 40,460 women are expected to die of breast cancer in the coming year, making the disease the second leading cause of cancer-related mortality among women (trailing only cancers of the lung and bronchus). However, thanks in part to recent advances in treatment, mortality rates associated with breast cancer have declined consistently since 1990.

Surgical resection and other treatments may particularly benefit patients whose disease is identified prior to metastasis; the 5-year survival rate for patients diagnosed with locoregionally advanced disease is 83%. However, women with distant metastases at diagnosis have a much poorer outlook, with a 5-year survival rate of only 26% and a median survival of approximately 2 years. Treatment of advanced disease may include first-line chemotherapy utilizing an anthracycline (eg, doxorubicin or epirubicin), antibody therapy, limited surgery, taxanes, and other cytotoxic agents. As complete responses are rare, these treatments are not generally employed as curative but in an effort to prolong life and provide symptom palliation.

Approximately two-thirds of all breast cancers are positive for expression of the estrogen receptor.For patients whose tumors are positive for this receptor or the progesterone receptor, the preferred first-line treatment comprises blockade of estradiol synthesis or hormone receptor activity using aromatase inhibitors or antiestrogen agents. Although endocrine therapies are useful and well-tolerated, most patients respond to this form of treatment for about 12-18 months before developing refractory disease. New therapies able to provide additional benefit to patients with hormone receptor-positive, antiestrogen-refractory, advanced and metastatic breast cancer are required.

ELIGIBILITY:
Inclusion Criteria:

* The patient has histologically or cytologically-confirmed invasive breast cancer, which at the time of study entry is either stage III (locally advanced) disease not amenable to curative therapy or stage IV disease. Histological confirmation of recurrent/metastatic disease is not required if clinical evidence of stage IV disease recurrence is available
* Tumors are positive for estrogen receptors (ER), progesterone receptors (PgR), or both (ie, 10% or more of infiltrating cancer cells exhibit nuclear staining for ER and/or PgR; positive biochemical test results are also acceptable)
* The patient has received prior antiestrogen therapy:

  1. With at least one antiestrogen agent (with or without ovarian suppression) administered for ≥ 3 months in the adjuvant or metastatic setting; and
  2. Experienced disease progression while on or within 12 months after receiving the last dose of endocrine therapy
* The patient is postmenopausal and/or meets at least one of the following criteria:

  1. Age ≥ 18 years with an intact uterus and amenorrhea for ≥ 12 months, with estradiol and/or follicle-stimulating hormone (FSH) values in the postmenopausal range
  2. History of bilateral oophorectomy
  3. History of bilateral salpingo-oophorectomy
  4. History of radiation castration and amenorrheic for ≥ 3 months
* The patient has fasting serum glucose < 120 mg/dL or below the ULN

Exclusion Criteria:

* The patient has received more than two regimens of prior chemotherapy in the metastatic (or locally advanced and inoperable breast cancer) and adjuvant setting
* The patient has poorly controlled diabetes mellitus. Patients with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range (fasting glucose at study entry < 120 mg/dL or below ULN) and that they are on a stable dietary and/or therapeutic regimen for this condition
* The patient is known to be positive for infection with the human immunodeficiency virus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2008-08; Primary Completion 2012-03 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - ImClone Investigational Site, Scottsdale, Arizona
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Westwood, Kansas
  - ImClone Investigational Site, Rochester, Minnesota
  - ImClone Investigational Site, Lebanon, New Hampshire
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, The Bronx, New York
  - ImClone Investigational Site, Columbus, Ohio
  - ImClone Investigational Site, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had progressive disease (PD) were considered to complete the study
Period: Overall Study
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Started | 62 | 31
Completed | 51 | 27
Not Completed | 11 | 4
Not completed — Adverse Event | 8 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Abnormal Lab Results | 0 | 2
Not completed — On treatment at cutoff date | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All randomized participants who were randomized regardless of actual treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab) | Total
Number analyzed (Participants) | 62 | 31 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 24 | 61
  >=65 years | 25 | 7 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 31 | 93
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 61 | 30 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 55 | 26 | 81
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization until date of objectively determined progressive disease (PD) or death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a ≥20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions unequivocal progression of non-target lesions. Participants without documentation of progression or death will be censored at the date of last tumor assessment. The PFS will be estimated following the Kaplan-Meier method.
Time Frame: From randomization up to 35.1 Months
Population: Intent-to-treat (ITT) population: All randomized participants who were randomized regardless of actual treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Number analyzed (Participants) | 62 | 31
months | 2.0 [1.9 to 3.4] | 3.1 [1.9 to 4.2]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) and Partial Response (PR) (Objective Response Rate [ORR])
Description: Best overall response of CR or PR was defined using RECIST v 1.0 criteria. CR was defined as the disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR was defined as ≥30% decrease in sum of longest diameter (SOD) of target lesions taking as reference the baseline sum diameter. PD was defined as ≥20% increase in SOD of target lesions and short axes of target lymph nodes, taking as reference the smallest sum of the longest diameters recorded since treatment started and an absolute increase in sum diameter of ≥5 mm; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. Percentage of participants=(number of participants with CR+PR/total number of participants)*100.
Time Frame: Randomization to PD up to 35.1 Months
Population: Intent-to-treat (ITT) population: All randomized participants who were randomized regardless of actual treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Number analyzed (Participants) | 62 | 31
percentage of participants | 1.6 [0.0 to 8.7] | 0 [0.0 to 11.2]

3. Secondary Outcome: 12-Month Survival Rate
Description: The 12-month survival rate is defined as the percentage of participants who have not died 12 months after the date of randomization.
Time Frame: From randomization to until the date of first documented date of death from any cause within 12 months, assessed up to 35.1 months
Population: Intent-to-treat (ITT) population: All randomized participants who receive any drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Number analyzed (Participants) | 62 | 31
percentage of participants | 15 [7.5 to 25.0] | 7.6 [1.9 to 18.7]

4. Secondary Outcome: Percentage of Participants With Complete Response (CR) and Partial Response (PR) or Stable Disease (SD) Disease Control Rate [DCR])
Description: DCR is defined as percentage of participants with CR, PR, or SD using RECIST v 1.0 criteria. CR: disappearance of all lesions, pathological lymph node reduction in short axis to <10 mm, and normalization of tumor marker levels of non-target lesions. PR: ≥30% decrease in SOD of target lesions taking as reference baseline sum diameter. PD: ≥20% increase in SOD of target lesions and short axes of target lymph nodes, taking as reference smallest sum of longest diameters recorded since treatment started and an absolute increase in sum diameter ≥5 mm; appearance of ≥1 new lesions and/or unequivocal progression of existing non-target lesions. SD: neither sufficient shrinkage to qualify for PR nor increase to qualify for PD. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. Percentage of participants=(number of participants with CR+PR+SD/total number of participants)*100.
Time Frame: Randomization to PD up to 35.1 Months
Population: Intent-to-treat (ITT) population: All randomized participants who were randomized regardless of actual treatment. Number of participants censored = 15 Cixutumumab + antiestrogen, 5 Cixutumumab only
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Number analyzed (Participants) | 62 | 31
percentage of participants | 40.3 [28.1 to 53.6] | 51.6 [33.1 to 69.8]

5. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) in National Cancer Institute Common Toxicity Criteria for AE's (NCI-CTCAE) Version 3.0 Criteria for Adverse Events (NCI-CTCAE)
Description: The NCI-CTCAE provides descriptive terminology for adverse event reporting. A grading (severity) scale is provided for each adverse event term. Severity will be graded as mild (grade 1), moderate (grade 2), severe (grade 3), or very severe (life threatening - grade 4). Clinically significant events were defined as serious and other non-serious adverse events related to study drug regardless of causality. A summary of serious and other non-serious adverse events is located in the Reported Adverse Event module.
Time Frame: Randomization to End of Study up to 36.5 Months
Population: Safety population: All participants who received actual treatment of any drug. There is a difference of 6 participants for treatment groups of IMC-A12 (Cixutumumab) + Antiestrogen and IMC-A12 (Cixutumumab) of ITT population and Safety population due to planned treatment (based on randomization) differed from actual treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Number analyzed (Participants) | 56 | 37
Participants
  Participants with any AE | 55 | 36
  Participants with SAE's | 16 | 11
  AE of greater than Grade 3 | 22 | 19
  AE with outcome of Death | 3 | 2
  Study drug-related AE | 48 | 31
  Study drug-related SAE's | 5 | 2
  Study drug-related AE of greater than Grade 3 | 10 | 7
  AE leading to discontinuation of any study drug | 6 | 1

6. Secondary Outcome: Changes in Circulating Tumor Cell Counts (CTS)
Time Frame: Approximately 24 months
Population: Zero participants analyzed. Circulating tumor cell counts were not collected for analysis.
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the interval between date of randomization and the date of death due to any cause. Participants who are alive at the time of study completion will be censored at the time the participants was last known to be alive.
Time Frame: From randomization up to 36.5 Months
Population: Intent-to-treat (ITT) population: All randomized participants who were randomized regardless of actual treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Number analyzed (Participants) | 62 | 31
months | 20.3 [11.5 to NA] — Below the level of detection, due to small survival data. | NA [17.8 to NA] — Below the level of detection, due to small survival data.

ADVERSE EVENTS:
Description: There is a difference of 6 participants for treatment groups of IMC-A12 (Cixutumumab) + Antiestrogen and IMC-A12 (Cixutumumab) of ITT population and Safety population due to planned treatment (based on randomization) differed from actual treatment.
Arm/Group | IMC-A12 (Cixutumumab) + Antiestrogen Therapy | IMC-A12 (Cixutumumab)
Serious Adverse Events (participants affected / at risk) | 16/56 | 11/37
Other Adverse Events (participants affected / at risk) | 55/56 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 (Cixutumumab) + Antiestrogen Therapy (N=56) | IMC-A12 (Cixutumumab) (N=37)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Disease progression (General disorders) | 2 (2) | 2 (2)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12 (Cixutumumab) + Antiestrogen Therapy (N=56) | IMC-A12 (Cixutumumab) (N=37)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Photopsia (Eye disorders) | 4 (4) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (11) | 4 (8)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 14 (16)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 18 (23) | 11 (11)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 10 (14) | 9 (12)
Asthenia (General disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 22 (32) | 20 (28)
Infusion related reaction (General disorders) | 4 (4) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 5 (5) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Thirst (General disorders) | 0 (0) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (8)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 24 (32) | 18 (26)
Anorexia (Metabolism and nutrition disorders) | 9 (10) | 10 (13)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (10) | 8 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (11) | 4 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2)
Dizziness (Nervous system disorders) | 8 (9) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (10)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (7)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 8 (10) | 4 (5)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
There is a difference of 6 participants for treatment groups of IMC-A12 (Cixutumumab) + Antiestrogen and IMC-A12 (Cixutumumab) of ITT population and Safety population due to planned treatment (based on randomization) differed from actual treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days